CLINICAL TRIAL: NCT02943798
Title: Optimization for the Treatment of Advanced Pulmonary Large Cell Neuroendocrine Carcinoma: a Prospective, Randomized, Open-label, Phase 2 Study
Brief Title: Optimization for the Treatment of Advanced Pulmonary Large Cell Neuroendocrine Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Zhou Zhen, Chief Physician, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chest003
Record Dates: First submitted 2016-10-22; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Large Cell Neuroendocrine Carcinoma
Keywords: Pulmonary Large Cell Neuroendocrine Carcinoma,chemotherapy
MeSH Terms: interventions — Etoposide; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Patients will be administered with etoposide plus carboplatin as first-line treatment.
  Interventions: Drug: etoposide plus carboplatin
- Group B (Experimental): Patients will be administered with paclitaxel plus carboplatin as first-line treatment.
  Interventions: Drug: Paclitaxel plus carboplatin

INTERVENTIONS:
Drug: etoposide plus carboplatin — etoposide is administered by venus with a dose of 100mg/m2 from day 1 to3, and carboplatin is administered by venus with a dose of AUC 5 on day 1 in a 21-day cycle.
  Other Names: VP-16
  Arms: Group A
Drug: Paclitaxel plus carboplatin — Paclitaxel is administered by venus with a dose of 175 mg/m2 from day 1 and carboplatin is administered by venus with a dose of AUC 5 on day 1 in a 21-day cycle.
  Other Names: Taxol
  Arms: Group B

SUMMARY:
The primary endpoint is to compare the PFS (progress-free survival ) of etoposide plus carboplatin with paclitaxel combined with carboplatin as first-line treatment for advanced pulmonary large cell neuroendocrine carcinoma.

DETAILED DESCRIPTION:
The primary endpoint is to compare the PFS (progress-free survival ) of etoposide plus carboplatin with paclitaxel combined with carboplatin as first-line treatment for advanced pulmonary large cell neuroendocrine carcinoma.

In addition, gene spectrum detection and Mini-PDX are applied for validation of pharmacodynamic.

Results of clinical trials and pharmacodynamic test will be analyzed to provide evidence for the precise treatment for LCNEC.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or IV pulmonary large-cell neuroendocrine carcinoma confirmed by histology or cytology
* Estimated life expectancy over 3 months
* Performance status 0,1,2
* Signed informed consent
* Adequate organ functions: absolute neutrophil count (ANC) over 1,500 cells/mm3 (1.5 x 109/L); platelet count over100,000/mm3 (100 x 109/L); serum creatinine < 2.5 mg/dL (221 mmol/L); serum AST or ALT <5.0 x upper limit of normal (ULN); serum total bilirubin <2.0 mg/dL (34 mmol/L)

Exclusion Criteria:

* History of chemotherapy or molecular targeted therapy
* Thoracic radical radiotherapy within 28 days of the initiation of study drug therapy except for palliative radiotherapy
* Use of any standard/experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy
* Prior history of malignancies other than non-small cell lung cancer (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for > or = to 1 year
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating
* Patient with concurrent medical or psychiatric illness which would, in the opinion of the investigator, prevent compliance with the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 6 months
  Interval from randomization to disease progression, or untolerated toxicity

SECONDARY OUTCOMES:
Tumor response | 2 months
  Percentage of complete response and partial response

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhou, MD, Study Chair — Shanghai Chest Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fasano M, Della Corte CM, Papaccio F, Ciardiello F, Morgillo F. Pulmonary Large-Cell Neuroendocrine Carcinoma: From Epidemiology to Therapy. J Thorac Oncol. 2015 Aug;10(8):1133-41. doi: 10.1097/JTO.0000000000000589. PMID 26039012